CLINICAL TRIAL: NCT05450432
Title: Long-Term Maintenance With Ketamine and Esketamine for Reduction of Suicide in High-Risk Patients With Depression
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000972
Record Dates: First submitted 2022-06-16; First posted 2022-07-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: depression; suicidal ideation
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Suicidal Ideation | interventions — Ketamine; Esketamine

STUDY DESIGN:
Intervention Model Description: A total of 100 participants will be enrolled in the study to receive intravenous ketamine and intranasal esketamine. Participants will be compared against matched historical control subjects identified through electronic medical records.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ketamine and Esketamine Treatment (Other): All study subjects will receive intravenous (IV) ketamine and intranasal (IN) esketamine treatment.
  Interventions: Drug: Ketamine; Drug: Esketamine

INTERVENTIONS:
Drug: Ketamine — Study participants will start treatment including two ketamine infusion visits per week during the acute phase, for up to eight ketamine infusion visits. Participants will then be transitioned to maintenance with intranasal esketamine.
Drug: Esketamine — After one month from the eighth ketamine infusion visit, participants will initiate weekly esketamine for 12 weeks, for a total of 13 esketamine treatments. The esketamine visits will happen as per standard of care at the clinic and as instructed by the SPRAVATO Risk Evaluation and Mitigation Strategy.

SUMMARY:
The study will consist of a 24-week-long trial examining outcomes in patients with Major Depressive Disorder and suicidal ideation who will receive intravenous (IV) ketamine and intranasal (IN) esketamine, compared to a large sample of matched historical controls. Patients will be recruited from an inpatient psychiatric unit. Eligible patients who provided informed consent will be enrolled in the study that will include a eight IV ketamine treatments, 13 esketamine treatment visits, seven long assessment visits, five short assessment visits, and daily surveys. The study will examine the feasibility, tolerability, and efficacy of repeated IV ketamine followed by esketamine, as well as predictors of treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient at a psychiatric unit (or MGH medical unit, awaiting transfer to psychiatry).
2. Male and female, 18-70 years of age, inclusive, at screening.
3. Diagnosis of MDD, single or recurrent, and currently experiencing a major depressive episode (MDE) at least eight weeks in duration, prior to screening, according to the criteria defined in the Diagnosis and Statistical manual of Mental Disorders, Fifth Edition (DSM-5). The diagnosis of MDD will be made by a site psychiatrist and supported by the Mini-International Neuropsychiatric Interview (MINI).
4. Suicidal ideation determined by a minimum score of 1 on item 12 of the QIDS-C assessment and based on admission to the inpatient unit for suicidal thoughts or behaviors.
5. In good general health, as ascertained by medical history. If needed to verify health status, the investigator may order/conduct physical examination (PE) (including measurement of supine and standing vital signs), clinical laboratory evaluations, or ECG.
6. A status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

1. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening); or 2. Childbearing potential, and meets the following criteria:

1. Childbearing potential, including women using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent.
2. Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test prior to receiving study treatment.
3. Willing and able to continuously use a method of birth control during the course of the study (implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence). The form of birth control will be documented at screening.

7. Access to a mobile phone or computer with internet connection. 8. Ability to read, understand and provide written and dated informed consent prior to screening.

9. Must have a provider to manage psychiatric medication, such as a psychiatrist, nurse practitioner, primary care physician, etc., either prior to admission or at discharge from the inpatient unit.

Exclusion Criteria:

1. Any history of previous treatment with IV ketamine.
2. Pregnant or breastfeeding.
3. Subject of childbearing potential who is not willing to use birth control during the study.
4. Unstable medical illness, i.e., severe liver or kidney disease, uncontrolled hypertension, uncontrolled hyperthyroidism
5. Current diagnosis of a moderate to severe substance use disorder (excluding mild or moderate alcohol or cannabis use disorder which will be permitted), within the last six months prior to screening based on DSM-5 criteria.
6. History of bipolar disorder, or any psychotic symptoms in the current or previous depressive episodes.
7. An Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within six months prior to screening (i.e., eating disorder, OCD, PTSD).
8. Currently receiving ECT treatment.
9. Currently receiving frequent or high dose benzodiazepines, opiates, barbiturates, or other CNS depressant medications, based on an increased risk of sedation in combination with ketamine.
10. Has dementia, delirium, amnestic, or any other primary cognitive disorder.
11. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results according to a licensed physician on the study staff.
12. Inability to consent to or comply with the study procedures.
13. Other medical issues:

    1. Hypertension, (SBP ≥160 mmHg or DBP ≥100 mHg) at Screening - untreated
    2. Recent myocardial infarction (within one year)
    3. Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system (CNS) disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention which, according to the screening done by a licensed physician, is deemed associated with significant injury to or malfunction of the CNS, or history of significant head trauma within the past 2 years
    4. Thyroid stimulating hormone (TSH) outside of the normal limits and clinically significant as determined by the Investigator.
    5. Any other clinically significant abnormal laboratory result (determined as such by the Investigator and/or medical monitor) at the time of the screening.
    6. Patients with diabetes mellitus fulfilling any of the following criteria:

1. Unstable diabetes mellitus defined as glycosylated hemoglobin (HbA1c) >8.5% at screening.

2. Admitted to hospital for treatment of diabetes mellitus or diabetes mellitus- related illness in the past 12 weeks.

g. Patients with a history of narrow angle glaucoma - untreated 14. Inability to comply with ketamine clinic safety procedures, including having reliable escorts to and from visits.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Retention | 24 weeks
  For examining the feasibility of treatment with ketamine and esketamine, descriptive analyses will be conducted to assess participants' retention across study visits.
Feasibility - Drop-out Rates | 24 weeks
  For examining the feasibility of treatment with ketamine and esketamine, descriptive analyses will be conducted to assess participants' drop-out rates across participation in the study.
Tolerability - Cognitive Function and Side Effects | Weeks 0, 1, 2, 3, 4, 8, and 12-24
  In regard to tolerability, the investigators will closely monitor cognitive functions and side effects during the administration of ketamine and esketamine.
Tolerability - Dosage of Treatment | Change between weeks 0, 4, 6, 8, 10, 12, 14, 16, 20, 22, and 24
  In regard to tolerability, the investigators will record the Necessary Clinical Adjustments (NCAs) for dosage of ketamine and esketamine treatments.
Tolerability - Frequency of Treatment | Change between weeks 0, 4, 6, 8, 10, 12, 14, 16, 20, 22, and 24
  In regard to tolerability, the investigators will record the Necessary Clinical Adjustments (NCAs) for the frequency of ketamine and esketamine administration.

SECONDARY OUTCOMES:
Efficacy - Treatment Response | Weeks 4, 8, and 12-24
  Descriptive analyses will be performed for percentage of responders (defined as 35% improvement on the QIDS-16) at the end of the IV ketamine acute phase, after the eighth ketamine infusion, and across the esketamine maintenance phase.
Efficacy - Trajectory of Suicidal Ideation | 24 weeks
  The change in participants' suicidal ideation will be examined over time and compared to historical controls.
Efficacy - Trajectory of Depression | 24 weeks
  The change in participants' depression will be examined over time and compared to historical controls.
Efficacy - Hospital Readmission Rates | 24 weeks
  The change in participants' hospital readmission rates will be examined over time and compared to historical controls.
Efficacy - Prevalence of Suicidal Behavior | 24 weeks
  The occurrence of suicidal behavior (gestures, attempts, and completed suicide) among participants will be examined over time and compared to historical controls.
Efficacy - Healthcare Utilization | 24 weeks
  The change in participants' healthcare utilization rates will be examined over time and compared to historical controls.

OTHER OUTCOMES:
Exploratory Aim - Predictors of Treatment Response | 24 weeks
  Exploratory aims will be examined, including predictors of treatment response (defined as 35% improvement in QIDS score) at the end of the acute and maintenance phases.
Exploratory Aim - Predictors of Suicidal Ideation Relapse | 24 weeks
  Exploratory aims will be examined, including predictors of suicidal ideation relapse (defined as SSI5>1) during time intervals between intravenous ketamine visits and during the esketamine maintenance phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share IPD.